CLINICAL TRIAL: NCT03576508
Title: A Two-Period Crossover Study to Compare the Systemic Exposure to Trans-Capsaicin and Cis-Capsaicin From an Intra-Articular Injection of CNTX-4975-05 (Trans-capsaicin for Injection) and Topical 8% Capsaicin Patch (Qutenza®) in Subjects With Painful Knee Osteoarthritis
Brief Title: A Study to Compare Levels of Capsaicin After Intra-Articular Injection and Topical Application in Patients With Painful Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CNTX-4975i-OA-102
Record Dates: First submitted 2018-06-11; First posted 2018-07-03 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Capsaicin; zucapsaicin; Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CNTX-4975-05 Intra-Articular (IA) Injection (Experimental): Receives IA injection into the most painful OA knee.
  Interventions: Drug: CNTX-4975-05; Drug: Lidocaine (without epinephrine)
- Topical 8% Capsaicin Patch (Active Comparator): Receives Capsaicin Patch on posterior rib cage.
  Interventions: Drug: Qutenza

INTERVENTIONS:
Drug: CNTX-4975-05 — 1 mg (2mL) IA injection
  Other Names: trans-capsaicin
  Arms: CNTX-4975-05 Intra-Articular (IA) Injection
Drug: Qutenza — 8% topical patch
  Other Names: cis-capsaicin
  Arms: Topical 8% Capsaicin Patch
Drug: Lidocaine (without epinephrine) — 15 mL IA injection of 2% lidocaine (without epinephrine)
  Arms: CNTX-4975-05 Intra-Articular (IA) Injection

SUMMARY:
This is a Phase 1b, open-label, two-period, randomized crossover study in adult male and female participants with painful knee osteoarthritis.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) between 18.0-35.0 kg/m^2
* Subject has moderate to severe painful osteoarthritis in one knee while walking (index knee); contralateral knee may or may not have osteoarthritis, pain should be none to mild in the non-index knee
* Confirmation of the OA of the index knee: American College of Rheumatology (ACR) diagnostic criteria
* Subject has intact skin at the location of the dosing sites (patch or injection)

Key Exclusion Criteria:

* Subject has any other form of arthritis, such as, but not limited to, rheumatoid arthritis, psoriatic arthritis, gout, systemic lupus erythematosus, etc.
* Subject has a dermatological condition that may contraindicate participation, including any compromise in skin integrity at the CNTX-4975-05 injection site or the Qutenza® skin application site, e.g., severe or cystic acne, psoriasis, eczema, atopic dermatitis, active or treated cancer, etc.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Capsaicin Pharmacokinetics - AUC0-t | Day 1 (pre-dose to 12 hours post-dose) and Day 8 (pre-dose to 12 hours post-dose)
  Single-dose systemic exposure to trans- and cis-capsaicin measured by AUC0-t.
Capsaicin Pharmacokinetics - AUC0-inf | Day 1 (pre-dose to 12 hours post-dose) and Day 8 (pre-dose to 12 hours post-dose)
  Single-dose systemic exposure to trans- and cis-capsaicin measured by AUC0-inf.
Capsaicin Pharmacokinetics - Cmax | Day 1 (pre-dose to 12 hours post-dose) and Day 8 (pre-dose to 12 hours post-dose)
  Single-dose systemic exposure to trans- and cis-capsaicin measured by Cmax.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) Assessment | Day 1 (pre-dose) or Day 8 (pre-dose) [cross over trial Qutenza® 8% patch or CNTX-4975-05 intra-articular (IA) knee injection], and Week 8 (follow-up)
  Change from baseline in KOOS of IA injected knees; 5-point Likert scale: 0 (no problems) to 4 (extreme problems); 5 subscales; each assessed separately
Incidence of treatment-emergent adverse events (TEAEs) (safety and tolerability) | Day 1 (post-dose), Day 8 (post-dose), and Week 8 (follow-up)
  Number of participants with TEAEs, which includes laboratory test variables
IA knee Lidocaine Systemic Pharmacokinetics - Concentration | Day 1 (pre-dose to 3 hours post-dose) or Day 8 (pre-dose to 3 hours post-dose) [Cross over trial Qutenza® 8% patch or CNTX-4975-05 IA knee injection]
  System exposure to lidocaine measured by plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Randall Stevens, MD, Study Chair — Centrexion Therapeutics
Locations (1):
- Well Pharma Medical Research, Corp, Miami, Florida, United States